CLINICAL TRIAL: NCT04794491
Title: A Phase 4 Multicenter, Open-label, Single-arm Study of Safety, Tolerability, Effectiveness and Treatment Optimization in Participants Switching From Xyrem to XYWAV for the Treatment of Narcolepsy
Brief Title: An Interventional Safety Switch Study (Segue Study) of XYWAV in Narcolepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JZP258-401
Record Dates: First submitted 2021-02-25; First posted 2021-03-12 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label Conversion and Treatment Optimization (Experimental): Conversion from Xyrem to XYWAV, maintaining the dose and regimen of any concomitant anticataplectics or stimulants unchanged throughout study.
  Interventions: Drug: JZP-258

INTERVENTIONS:
Drug: JZP-258 — Maximum nightly dosage of 9 grams, administered once, twice or thrice nightly, with no single dose > 6 g
  Other Names: XYWAV

SUMMARY:
The rationale for the interventional, open-label, single-arm design of JZP258-401 is to evaluate the clinical experience in participants with narcolepsy transitioning treatment from Xyrem to XYWAV.

ELIGIBILITY:
Inclusion Criteria:

Age

1. Participant must be 18 to 80 years of age (inclusive), at the time of signing the informed consent. Type of Participant and Disease Characteristics
2. Participants who have a primary diagnosis of Type 1 or Type 2 narcolepsy that meets ICSD-3 criteria or DSM-5 criteria (Ruoff and Rye 2016), and are being currently treated with Xyrem, with or without additional anticataplectics or stimulants.
3. Participants who have been taking Xyrem (with or without additional anticataplectics or stimulants eg, TCA, SNRI, SSRI, atomoxetine) in a stable dose and regimen for at least two months prior to screening, with evidence of clinical improvement on their current regimen, per the investigator's judgement. Only Xyrem will be substituted with XYWAV, with dose and regimen of any concomitant anticataplectics or stimulants remaining unchanged throughout the study.

   Sex and Contraceptive/Barrier Requirements
4. Participant is male or female

   * A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

     * Is a woman of non-childbearing potential (WONCBP) as defined in Appendix 3 OR
     * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of < 1% per year), preferably with low user dependency, as described in Appendix 3, during the study Intervention period and for at least 7 days after the last dose of study intervention. The investigator should evaluate the potential for contraceptive method failure (eg, noncompliance, recently initiated) in relationship to the first dose of study intervention.
   * A WOCBP must have a negative highly sensitive pregnancy test (serum) during screening.
   * The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

   Informed Consent
5. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

Medical Conditions

1. Have a diagnosis of narcolepsy, secondary to another medical condition (eg, central nervous system injury or lesion)
2. Are currently prescribed a Xyrem regimen exceeding a dose of 9 grams nightly, or any single dose in excess of 6 grams.
3. Have been diagnosed with restless leg syndrome (RLS) requiring treatment other than iron supplements
4. Exhibit succinic semi-aldehyde dehydrogenase deficiency (SSADH)
5. Have uncontrolled hypothyroidism
6. Have a history of seizures, excluding early childhood non-pathological febrile seizures
7. Have a history of head trauma associated with loss of consciousness in the past 5 years, or if the event occurred more than 5 years prior to screening and the participant experiences sequelae due to the event
8. Show evidence of untreated or inadequately treated sleep-disordered breathing including:

   1. Presence of clinically significant and untreated obstructive or central sleep apnea (as determined by the investigator or documented previously); or one of the following:
   2. Apnea index (AI) >10 if on Obstructive Sleep Apnea (OSA) treatment or untreated, or
   3. Clinically significant hypoventilation, or
   4. Noncompliance with primary OSA therapy Note: "Non-compliance" is defined as positive airway pressure use of <4 hours per night on <70% of nights (<5 of 7 nights/week) per historical report (with investigator concurrence) of use of an oral appliance on <70% of nights (≥5 of 7 nights/week), or receipt of an effective surgical intervention for OSA symptoms.
9. Experience parasomnias (eg, sleep walking, REM Sleep Behavior Disorder, etc.) considered by the investigator to negatively impact the conduct of the study. Parasomnia events associated with physical injury to the participant (or others) shall be discussed with the sponsor Medical Monitor.
10. Meet criteria for current major depression based on clinical interview
11. Have any clinically relevant medical, behavioral, or psychiatric disorder (other than narcolepsy) that is associated with excessive sleepiness
12. Have a history or presence of bipolar disorder, bipolar related disorders, schizophrenia, schizophrenia spectrum disorders, or other psychotic disorders according to DSM-5 criteria
13. Have a history or presence of any unstable or clinically significant medical condition, behavioral or psychiatric disorder (including active suicidal ideation), or history or presence of another neurological disorder or surgical history that might affect the participant's safety and/or interfere with the conduct of the study, in the opinion of the investigator
14. Display relevant suicidality as indicated by Columbia Suicide Severity Rating Scale (C-SSRS) evaluation at screening
15. Display moderate to severe depression as indicated by the Participant Health Questionnaire - 9 (PHQ-9) at screening
16. Are a female participant who is pregnant or breastfeeding

    Prior/Concomitant Therapy
17. Have undergone treatment with any prohibited central nervous system (CNS) agents, including but not limited to benzodiazepines, non-benzodiazepine anxiolytics/ hypnotics/sedatives, neuroleptics, opioids, barbiturates, phenytoin, ethosuximide, or MCT inhibitors, eg, diclofenac, valproate, ibuprofen, within 2 weeks prior to enrollment. Discontinuation for the purpose of study enrollment is permitted only if considered safe by the investigator and approved by the Medical Monitors.

    Prior/Concurrent Clinical Study Experience
18. Received any other investigational drug within 30 days or five half-lives (whichever is longer) prior to screening, or plan to use an investigational drug (other than the study intervention) during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Wright Clinical Research, LLC, Alabaster, Alabama
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Pulmonary Associates of the Southeast, PC, Birmingham, Alabama
  - Santa Monica Clinical Trials, Los Angeles, California
  - Southern California Institute For Respiratory Diseases, Inc./ Tower Sleep Medicine, Los Angeles, California
  - Southern California Institute For Respiratory Diseases, Inc., Los Angeles, California
  - Stanford University- Sleep Medicine, Redwood City, California
  - SDS Clinical Trials, Inc, Santa Ana, California
  - Delta Waves, Inc., Colorado Springs, Colorado
  - Pulmonary Disease Specialists, PA d/b/a PDS Research, Kissimmee, Florida
  - Clinical Research of West Florida, Inc, Tampa, Florida
  - Florida Pediatric Research Institute, LLC, Winter Park, Florida
  - Sleep Practitioners LLC, Macon, Georgia
  - Clinical Research Institute, Stockbridge, Georgia
  - The Center for Sleep & Wake Disorders, Chevy Chase, Maryland
  - WMed Center for Clinical Research, Kalamazoo, Michigan
  - Minnesota Lung Center, Edina, Minnesota
  - Clayton Sleep Institute, LLC, St Louis, Missouri
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Intrepid Research LLC, Cincinnati, Ohio
  - Cleveland Clinic, Sleep Disorders Center, Cleveland, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Geisinger Clinic, Danville, Pennsylvania
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - Medical University of South Carolina, Department of Psychiatry and Behavioral Sciences, North Charleston, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Macfadden W, Leary EB, Fuller DS, Kirby MT, Roy A. Effectiveness and optimization of low-sodium oxybate in participants with narcolepsy switching from a high-sodium oxybate: data from the Substitution of Equal Grams of Uninterrupted Xyrem to Xywav study. J Clin Sleep Med. 2024 Sep 1;20(9):1467-1477. doi: 10.5664/jcsm.11182. PMID 38652499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 62 participants were enrolled in trial sites across the United States.
Groups:
- Overall: Participants received JZP258 (XYWAV) at a maximum nightly dosage of 9 g administered orally 1 to 3 times nightly, with no single dose exceeding 6 g.
Period: Overall Study
Arm/Group | Overall
Started | 62
Baseline Period | 62
Intervention (XYWAV) Period | 60
Safety Follow-Up Period | 59
Completed | 54
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Alcohol or Urine Drug Screen Result Is Positive | 4
Not completed — Noncompliance With Study Intervention | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the Safety Analysis Set, which included all participants in the Enrolled Analysis set who received at least 1 dose of Xyrem after providing informed consent.
Arm/Group | Overall
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (15.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 54
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Weekly Rate of Cataplexy Attacks
Description: Mean weekly rate of cataplexy attack = (total number of cataplexy attacks reported during the period/number of days during the period where a diary was completed) x 7.
Time Frame: Baseline to Week 8
Population: The weekly rate of cataplexy attacks was assessed using the XYWAV Efficacy Analysis Set, which included all participants in the XYWAV Safety Analysis Set who finished the course of study. Includes Narcolepsy type 1 participants with a mean weekly rate of cataplexy attack at both the first 7 days of the baseline period and the week 8 visit.
Measure: Mean (Standard Deviation); unit: cataplexy attacks per week
Arm/Group | Overall
Number analyzed (Participants) | 24
cataplexy attacks per week | 0.98 (4.1222)

2. Other Pre Specified Outcome: Change in the Nausea Visual Analog Scale (NVAS)
Description: Tolerability associated with Xyrem and XYWAV was measured based on an NVAS assessment administered electronically. NVAS was captured daily during the last 7 days of the Baseline (Xyrem-stable dose and regimen) period and the last 7 days of the Intervention period (on XYWAV) prior to the ET visit or prior to the E/D visit, if possible. For participants with at least one day of NVAS data, the NVAS for that week was the average daily score from days with non-missing data within the week, then multiplied by 7. The NVAS ranges 0-100 mm, with higher scores representing more severe/intense nausea.
Time Frame: Baseline to Week 8
Population: NVAS was assessed using the XYWAV Efficacy Analysis Set, which included all participants in the XYWAV Safety Analysis Set who finished the course of study. Includes participants with a baseline value and a post-baseline value at the end of treatment (ET) or early discontinuation ( E/D).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall
Number analyzed (Participants) | 47
score on a scale | 3.13 (29.089)

3. Other Pre Specified Outcome: Number of Participants With Patient Global Impression of Change (PGIc) Values
Description: The PGIc is a 7-point Likert-type rating based on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). PGIc values were measured at the ET or E/D, as applicable.
Time Frame: Week 8
Population: PGIC was assessed using the XYWAV Efficacy Analysis Set, which included all participants in the XYWAV Safety Analysis Set who finished the course of study. Includes participants who have at least one PGIc assessment performed at the end of the intervention period or early discontinuation (E/D) visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall
Number analyzed (Participants) | 51
Participants
  Very Much Improved | 1
  Much Improved | 9
  Minimally Improved | 12
  No Change | 26
  Minimally Worse | 3
  Much Worse | 0
  Very Much Worse | 0

4. Other Pre Specified Outcome: Change in Epworth Sleepiness Scale (ESS)
Description: The ESS questionnaire included a set of 8 questions regarding how likely the participant would be to doze off or fall asleep in different situations. The ESS measures EDS or average sleep propensity in daily life. Responses range from 0 = would never doze (better outcome) to 3 = high chance of dozing (worse outcome). Changes in ESS scores were assessed between the Baseline period and ET or E/D, as applicable
Time Frame: Baseline to Week 8
Population: ESS was assessed using the XYWAV Efficacy Analysis Set, which included all participants in the XYWAV Safety Analysis Set who finished the course of study. Includes participants with Epworth Sleeping Scale assessments at both Baseline and ET or E/D visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall
Number analyzed (Participants) | 50
units on a scale | -0.6 (2.33)

5. Other Pre Specified Outcome: Time to Achieve Optimized Dose and Regimen
Description: Defined as the time from the first dose and regimen to the optimized dose and regimen of XYWAV, where the optimized dose and regimen indicates the final dose and regimen that remains unchanged throughout the remainder of the Intervention period.
Time Frame: Baseline to Week 8
Population: The time to achieve an optimized dose and regimen was assessed using the XYWAV Efficacy Analysis Set, which included all participants in the XYWAV Safety Analysis Set who finished the course of study.
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Overall
Number analyzed (Participants) | 54
day | 2.6 (4.90)

6. Other Pre Specified Outcome: Number of Changes From the First Dose and Regimen to Optimized Dose and Regimen
Description: The amount of times the dose and regimen were changed before an optimized dose and regimen were achieved.
Time Frame: Baseline to Week 8
Population: The number of changes from the first dose and regimen to the optimized was assessed using the XYWAV Efficacy Analysis Set, which included all participants in the XYWAV Safety Analysis Set who finished the course of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall
Number analyzed (Participants) | 54
Participants
  Never Changed | 48
  Changed Once | 6
  Changed Twice | 0
  Changed More than Twice | 0

7. Other Pre Specified Outcome: Number of Participants Dosing Fasted Versus Dosing Without Consideration of Food
Description: Once the participant reached an optimized dose and regimen, the investigator could decide to instruct the participant to dose without regard to food.
Time Frame: Baseline to Week 8
Population: The number of participants who dosed fasted versus without food consideration was assessed using the XYWAV Efficacy Analysis Set, which included all participants in the XYWAV Safety Analysis Set who finished the course of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall
Number analyzed (Participants) | 54
Participants
  Dosing Fasted | 53
  Dosing without Food Consideration | 1

8. Other Pre Specified Outcome: Duration of Time Between the Last Meal Relative to Dosing
Description: The difference between the time of day that participants ate their last meal and the time of day participants take their first dose.
Time Frame: Baseline to Week 8
Population: The duration of time between the last meal and dosing was assessed using the XYWAV Efficacy Analysis Set, which included all participants in the XYWAV Safety Analysis Set who finished the course of study.
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | Overall
Number analyzed (Participants) | 54
minute | 113.7 (313.31)

9. Other Pre Specified Outcome: Characterization of Meals Relative to Dosing
Description: Types of meals consumed before dosing.
Time Frame: Baseline to Week 8
Population: Characterization of meals was assessed using the XYWAV Efficacy Analysis Set, which included all participants in the XYWAV Safety Analysis Set who finished the course of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall
Number analyzed (Participants) | 54
Participants
  Regular Meal | 54
  Snack | 45
  Beverage Other than Water | 19

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event (TEAE) data were collected from up to 30 days before Day 1 up to week 10 + 3 days.
Description: A TEAE is defined as an AE that either began or worsened after administration of the first dose of study intervention (XYWAV) to End of Treatment Period (prior to the Safety Follow-up Period). Adverse events were assessed using the XYWAV Safety Analysis set, which included all participants in the Safety Analysis Set who received at least 1 dose of XYWAV.
Groups:
- Overall: Overall XYWAV safety analysis set.
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 2/60
Other Adverse Events (participants affected / at risk) | 18/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=60)
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=60)
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Oedema peripheral (General disorders) | 1
COVID-19 (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Sedation complication (Injury, poisoning and procedural complications) | 1
Urobilinogen urine increased (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Initial insomnia (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Urine abnormality (Renal and urinary disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT04794491/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT04794491/SAP_001.pdf